CLINICAL TRIAL: NCT04902560
Title: Overall Patient Care in a Montpelier Sexual Health Center (CeGIDD). Response Rate to Ceftriaxone 1g IM in Gonorrhoea : a French Retrospective Monocentric Study
Brief Title: Response Rate to Ceftriaxone 1g IM in Gonorrhoea : a French Retrospective Monocentric Study
Acronym: GONOCEF
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0301
Record Dates: First submitted 2021-05-18; First posted 2021-05-26 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Gonorrhea
Keywords: Neisseria gonorrhoea; Ceftriaxone; Treatment
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sexual health centers (CeGIDD, in France) manage the majority of STI in France, especially gonorrhea.

Patients wanting STI screening can consult either they are symptomatic or not.

If they are symptomatic, they can be treated immediately. If they are not symptomatic, they must come back seven days after in order to get their results and to be treated if necessary.

Before any treatment for gonorrhea, subjects should be sampled for bacterial culture in order to perform AMR surveillance.

After every treatment for gonorrhea, subjects should realized a test of cure (TOC) according to current recommandation.

Response rate to ceftriaxone 1g IM for treating gonorrhea has never been evaluated in France while being used widely over the past months.

Compliance to current recommandation at CeGIDD Montpellier has never been evaluated.

This study will assess the response rate to ceftriaxone 1g IM as gonorrhea treatment by realizing a test of cure 14 days after each treatment.

ELIGIBILITY:
Inclusion criteria:

* Aged more than 18 years old
* Non-opposition form given to the subject
* Having at least one exam positive for Gonorrhoea (PCR or Culture), realised in CeGIDD de Montpellier

Exclusion criteria:

- patient's refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient Having at least one exam positive for Gonorrhoea (PCR or Culture), realised in CeGIDD de Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Response rate to Ceftriaxone 1g IM in Gonorrhoea. | day 1
  Evaluated by a test of cure (TOC) which must be negative 15 days after the subject received the treatment (ceftriaxone).

SECONDARY OUTCOMES:
Adverse drug reaction rates | day 1
  Any adverse effect after treatment will be notified (digestive disorder, headache, phototoxicity, allergic reaction, local reaction at the site of injection…)
Concordance rate with positive PCR | day 1
  Before getting the treatment, all patients should have been sampled for bacterial culture according to current recommendation. Respect of the recommendation will be assessed by this outcome.
Resistance rate to ceftriaxone and AMR description. | day 1
  This measure will be assessed via bacterial cultures
Rate of untreated patient despite having a positive test for gonorrhea (lost to follow-up) | day 1
  Patient compliance may be lacking in sexual health center and non-compliance participate in STI spreading.
  Subject not looking for their results after being tested positive for gonorrhea will be notified by phone call. The necessity of calling the patient will be notified in the study.
  If the subject does not attend the medical consultation for treatment, he will be consider as lost to follow-up.
Rate of realized TOC | day 1
  Test of cure (TOC) is a PCR test realized at the previous positive site of contamination, approximately 14 days after treatment, in order to confirm the efficacity of treatment.
Rate of time before realizing the TOC. | day 1
  Sensibility and Specifity may differ depending on the time between treatment and the TOC.

CONTACTS AND LOCATIONS:
Overall Officials: Du Thanh Aurelie, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC